CLINICAL TRIAL: NCT05989906
Title: Feasibility of a Sprint Interval Training Program During Inpatient Spinal Cord Injury Rehabilitation: A Pilot Randomized Controlled Trial
Brief Title: Feasibility of a Sprint Interval Training Program During Inpatient Spinal Cord Injury Rehabilitation
Acronym: SIT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Deborah Crane, Associate Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00017002
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries
Keywords: Exercise; Mental Health; Feasibility; Inpatient Rehabilitation Unit; Sprint Interval Training
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity; Psychological Well-Being | interventions — High-Intensity Interval Training; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four treatment conditions:
  * Usual care
  * Sprint Interval Training
  * SIT + Home Ergometer
  * SIT + Home Ergometer + Motivational Interviewing
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research study assistant collecting self-report outcomes and Principal Investigators will be masked to participant's study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Usual Care (Active Comparator): Participant will take part in the usual care during inpatient rehabilitation
  Interventions: Behavioral: Usual Care
- Spring Interval Training (SIT) (Experimental): Participant will take part in SIT approximately three times per week during inpatient rehabilitation.
  Interventions: Behavioral: Sprint Interval Training (SIT)
- SIT + ERGO (Experimental): Participant will take part in SIT approximately three times per week during inpatient rehabilitation. In addition, participant will be provided with an consumer grade ergometer for home use.
  Interventions: Behavioral: Sprint Interval Training (SIT); Behavioral: Home Ergometer (ERGO)
- SIT + ERGO + MI (Experimental): Participant will take part in SIT approximately three times per week during inpatient rehabilitation. In addition, participant will be provided with an consumer grade ergometer for home use. The participant will receive Motivational Interviewing sessions with a rehab psychologist one time per week (approximately 4 sessions) during inpatient rehabilitation and one time per month for six months after discharge from the hospital
  Interventions: Behavioral: Sprint Interval Training (SIT); Behavioral: Home Ergometer (ERGO); Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Sprint Interval Training (SIT) — Participants will undergo 1:1 therapist supervised SIT for 10 minutes per day, three times per week during IPR using a Monark 881 arm crank ergometer.
  Arms: SIT + ERGO; SIT + ERGO + MI; Spring Interval Training (SIT)
Behavioral: Usual Care — Participants will have the opportunity to participate in optional group endurance exercise classes two to three times a week.
  Arms: Usual Care
Behavioral: Home Ergometer (ERGO) — Participants complete the SIT intervention during IPR and be provided with a consumer-grade ergometer. Study staff will train the participants in the set-up and use of the home ergometer prior to discharge and arrange for take home or delivery.
  Arms: SIT + ERGO; SIT + ERGO + MI
Behavioral: Motivational Interviewing (MI) — Participants complete the SIT intervention during IPR and be provided with a consumer-grade ergometer. Study staff will train the participants in the set-up and use of the home ergometer prior to discharge and arrange for take home or delivery. These participants will also receive weekly Motivational Interviewing (MI) counseling sessions during IPR plus six post-discharge MI sessions delivered via telehealth to be held over six months.
  Arms: SIT + ERGO + MI

SUMMARY:
This study will assess the feasibility and efficacy of 3 treatments to increase physical activity during and after inpatient rehabilitation (IPR) for new spinal cord injuries:

1. Program of sprint interval training (SIT) on an arm crank ergometer during IPR
2. SIT + Provision of an arm ergometer (ERGO) for home use
3. SIT + ERGO for home use + Motivational interviewing to increase adherence to exercise during and after IPR.

The primary outcome is minutes per week of moderate to vigorous physical activity at 6 months after IPR discharge. Secondary outcomes include peak power on the 6-Minute Arm Test at IPR discharge and self-reported physical activity, depression, fatigue, pain, community participation, and quality of life at 6 months after IPR discharge. The investigators will obtain data on feasibility, acceptability, and perceived benefits of the treatments from stakeholders. The results of this pilot study will inform the design of a larger randomized trial.

DETAILED DESCRIPTION:
Description of the Sprint Interval Training Condition

The SIT treatment procedures will parallel the procedures used in the successful comparative effectiveness trial of SIT versus Moderate Intensity Continuous Training (MICT) during IPR in Canada.

SIT participants will be trained to use an ergometer on a Monark 881 mechanically braked arm ergometer purchased for the study. The Monark will be mounted on a rolling table designed for this purpose, so training can take place in patient rooms or in one of several small therapy rooms adjacent to the inpatient rehabilitation unit. Sessions will begin with the physical or occupational therapist showing the participant the RPE scale (Borg 6-20) posted behind the ergometer and instructing the participant in how to report perceived exertion during each session. The therapist will position the ergometer axle at shoulder height and close enough to the participant to maintain slight elbow flexion. They will attach the heart rate monitor, validate initial recordings, assess resting RPE, and record resting HR and blood pressure. They will have the participant begin a two-minute warm-up at a self-selected speed and zero resistance followed by three 20-second intervals of all-out effort interspersed by 120 seconds of active recovery at zero resistance. During each interval, participants will be instructed to achieve a cadence of approximately 100 revolutions per minute for persons with paraplegia and approximately 85 revolutions per minute for people with tetraplegia. The therapist will adjust ergometer resistance as needed to maintain RPE ratings between 15-17. Rating of perceived exertion is a valid method to prescribe interval exercise intensity and preferable to HR. Heart rate will be recorded continuously and averaged over the entire training session excluding the warm-up and recovery periods. RPE will be measured at the end of each sprint interval training session. To accommodate training adaptation over time, the resistance on the ergometer will be increased to maintain a peripheral RPE of 16. SIT training was well-tolerated and safe in the prior IPR trial as well as in several post-acute SCI studies. Hypotension is a potential adverse event in this setting, especially immediately post-exercise. Thus, sessions will include blood pressure monitoring and surveillance for symptoms of hypotension during and after the exercise session. Adverse events will be reported to the research team for review by the DSMB. SIT training will take place approximately 3 times per week.

Description of the Home Arm Ergometer Condition

Participants randomized to receive ERGO will also take part in SIT approximately 3 times per week. Participants will undergo at least one SIT session on the consumer grade ergometer under supervision of the physical or occupational therapist. The therapist/team will demonstrate all the features of the device set up, use, and resistance adjustment to the patient and caregiver (if available). The therapist/team will problem-solve barriers to home use prior to discharge and contact the patient soon after discharge to help resolve additional problems that may have emerged. The patient will be sent home with an exercise log-sheet like the one used during IPR to guide continued training. Prior to discharge the study team will arrange to have the ergometer given to or shipped to the participant's discharge residence.

The investigators plan to give participants randomized to ERGO a consumer grade tabletop ergometer. Study staff will also provide ace bandages or specialized exercise gloves for patients with tetraplegia who cannot grip the ergometer handles.

Description of the Motivational Interviewing Condition

The motivational interviewing (MI) condition participants will take part in SIT approximately 3 times per week and be provided an ERGO for home use. In addition, participants will receive MI. The sessions will use a MI counseling style consisting of strategic use of open questions, reflections, affirmations, summaries, and information sharing. MI is a widely used, evidence-based counseling approach with evidence of efficacy across many different health behaviors including exercise promotion. The sessions will also include evidence-based content and behavior change principles such as goal setting, activity monitoring, feedback, and identification of barriers and facilitators. This content has been adapted for people with SCI from an unusually successful and highly replicated lifestyle intervention (the Diabetes Prevention Program (DPP)). The investigators will include 10 DPP modules on values and goals, self-monitoring, exercise safety, problem-solving I, relapse prevention, activity cues, problem-solving II, professional help, dealing with negative thoughts, and staying motivated. Participants will receive approximately four weekly 30-minute in-person counseling sessions during IPR and six monthly telehealth sessions during the post-discharge period provided by Dr. Bombardier, an expert in MI and exercise promotion.

Description of the Usual Care Control Condition

Study design includes a control group because our aims include preliminary efficacy as well as feasibility. The investigators chose Usual Care as the control group over other control group options, such as traditional moderate intensity aerobic conditioning in order to know whether the treatment components are potentially more effective than current standard of care. Also, traditional aerobic conditioning (30-45 minute sessions 3 times per week) is not a current component of IPR in the U.S. and is likely not feasible. All patients, including those assigned to usual care, may participate in optional group endurance exercise classes at the end of the day 2-3 times per week. Endurance group classes include moderate intensity continuous aerobic training using any equipment appropriate to the patient's level and severity of injury, as determined by the treating physical therapist.

Data Collection and Measurement Techniques There will be three assessment points: baseline, within the week prior to end of treatment/discharge from IPR, and at 6 months post discharge from IPR. All outcome assessments will be conducted by a trained and supervised research assistant who will be kept unaware of the participants treatment condition. Patient reported outcomes will be assessed via in-person structured interviews for baseline and discharge and via Zoom or telephone for 6-month assessments. A 6-MAT (6 minute arm test) will be done on an arm ergometer around the time of the baseline survey and repeated within one week prior to discharge from IPR. Participants will be asked to wear an Actigraph activity monitor for 1 week approximately 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with SCI
2. SCI below C2
3. AIS A-C
4. aged 18-65
5. undergoing acute IPR for SCI at Harborview Medical Center
6. Able to use an arm ergometer

Exclusion Criteria:

1. poorly controlled type II diabetes
2. unstable cardiovascular disease
3. shoulder injury
4. any other medical condition that would preclude safe participation in study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Total physical activity (vector magnitude) per week | 7 day assessment (at 6 month timepoint)
  To compare the effect sizes (Cohen's d) of each of the three treatment conditions: (1) SIT alone, (2) SIT+ERGO, and (3) SIT+ERGO+MI relative to usual care on the primary outcome, total physical activity (vector magnitude) per week at 6 months post discharge measured by an Actigraph GT3X worn on the non-dominant wrist for 7 days.
Percentage of participants that complete at least six Sprint Interval Training (SIT) sessions | Treatment Completion (week 3)
  Investigators will assess the total number and percentage of participants that complete at least six SIT sessions, the minimum number of SIT sessions associated with a significant increase in physical capacity among SCI participants.
Total number of Ergometer (ERGO) sessions that participants complete between treatment completion and 6 month follow up | 6 Month Follow Up (week 24)
  Among patients who received a home ergometer, the investigators will assess how many sessions of SIT the participants completed between treatment completion (in hospital) and the 6-month timepoint.
Percentage of participants that adhere to Sprint Interval Training sessions and received Motivational Interviewing (MI) sessions | 6 Month Follow Up (week 24)
  Investigators will assess the total number and percentage of participants that completed at least 75% of the Sprint Interval Training sessions among participants that received Motivational Interviewing.

SECONDARY OUTCOMES:
Adverse Events (Safety) | At the end of each Sprint Interval Training (SIT) session during weeks 0-4 of the study and at the end of the 6-minute arms tests (weeks 0-4)
  The investigators will ask participants at the end of each Sprint Interval Training (SIT) session, "Have you experienced any negative effects from today's training or as a result of participating in the study?" (Yes/No). If a participant responds 'Yes', investigators will ask for more details and will report this information to the Principal Investigators.
Acceptability | Treatment Completion (week 4), 6 Month Follow Up (week 24)
  The investigators will assess overall improvement on the Benefit, Satisfaction, and Willingness to Continue survey from Treatment Completion to 6 Month Follow Up. There are three questions:
  "Have you had any benefit from your treatment?" (Yes/No) "Taking all things into account, are you satisfied with your treatment?" (Yes/No) "Would you be willing to continue treatment with this therapy (Yes/No). Total scores range from 0-3 and greater total scores indicate greater satisfaction with treatment.
Peak power on the 6-Minute Arm Test (6-MAT) | Self-reported physical exertion at the end of 6 minutes of physical exercise on the arm ergometer at Baseline (week 0) and at Treatment Completion (week 4)
  Peak exertion on the 6-minute arm test measured by a physical therapist assisting the participant with the exercise. Self-reported scores range from 6-20, and higher scores indicate greater physical exertion.
Leisure Time Physical Activity (LTPA) | Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported mild to vigorous physical activity in the past week, reported as minutes per week and number of days per week of mild to vigorous physical activity. Greater total minutes and total days indicate more physical activity.
Patient Health Questionnaire (PHQ-9) | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported depression in the past week measured using a 9-item validated survey. Responses range from '0' (not at all) to '4' (nearly every day). Total scores range from 0-36 and higher total scores indicate worse depression.
Generalized Anxiety Disorder (GAD-7) | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported anxiety in the past week measured using a 7 item validated survey. Responses range from '0' (not at all) to '4' (nearly every day). Total scores range from 0-36 and higher total scores indicate worse anxiety.
Patient Reported Outcome Measures Information System (PROMIS) Fatigue Short Form | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported fatigue measured using a 4-item validated survey. Responses range from '0' (not at all) to '4' (very much). Total scores range from 0-16, with higher scores indicating worse fatigue.
Numerical Rating Scale (NRS) of Worst/Average Pain | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported worst and average pain in the past 7 days, rated from '0' (no pain) to '10' (pain as bad as you can imagine)
Wheelchair Users Shoulder Pain Inventory (WUSPI) | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported shoulder pain in the past week measured on a 10-point Likert scale from '0' (no pain) to '10' (worst pain ever experienced). Total scores range from 0-150 with greater total scores indicating greater pain.
Physical Activity Enjoyment Scale (PACES) | Within 5 minutes after each Sprint Interval Training session during first 3 weeks of study (weeks 0-3)
  Self-reported exercise enjoyment measured on a 7-point likert scale ranging from '0' (I hate it) to '7' (I enjoy it). Total scores range from 0-7 with greater scores indicating greater exercise enjoyment.
Spinal Cord Injury Exercise Self-Efficacy | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported exercise self-efficacy measured on a 4-point Likert scale from '0' (not true at all) to '4' (always true). Total scores range from 0-40, with greater scores indicating greater sense of self-efficacy.
SCI Quality of Life | Baseline (week 0), Treatment Completion (week 4), 6 Month Follow Up (week 24)
  Self-reported quality of life measured on a 10-point Likert scale using the International SCI Data Sets Quality of Life Basic Data sets survey, which has a 10-point Likert scale from '0' (Completely dissatisfied) to '10' (Completely satisfied). Total scores range from 0-30 with greater total scores indicating higher quality of life.
Oral Symbol Digit Modalities Test (SDMT) | Baseline (week 0), Treatment Completion (week 4)
  Brief neuropsychological assessment to measure cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Crane, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No